CLINICAL TRIAL: NCT06877624
Title: A Randomized, Open-Label, Single Dose, Cross-Over Study to Evaluate the Pharmacokinetics of Three QRL-101 Formulations in a Fasted Condition or in the Presence of a High Fat Meal in Healthy Participants
Brief Title: A Study Evaluating the Pharmacokinetics of Three QRL-101 Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QurAlis Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QRL-101-06
Record Dates: First submitted 2025-03-05; First posted 2025-03-14 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, open-label, single-dose, cross-over study to evaluate the pharmacokinetics of 3 QRL-101 formulations in a fasted condition or in the presence of a high-fat meal in healthy participants.
Who Masked: Participant, Investigator
Masking Description: A participant and investigator-blinded, randomized, open-label, single-dose, cross-over design will be used to minimize bias in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment Sequence 1 (Formulation 1, 2, and 3) (Experimental): Participants randomized to Treatment Sequence 1 will receive Formulation 1 in the fasted condition in Treatment Period 1, followed by Formulation 1, 2, and 3 in the presence of a high-fat meal in Treatment Periods 2 through 4, respectively.
  Interventions: Drug: QRL-101
- Treatment Sequence 2 (Formulation 2, 3, and 1) (Experimental): Participants randomized to Treatment Sequence 2 will receive Formulation 2 in the fasted condition in Treatment Period 1, followed by Formulation 2, 3, and 1 in the presence of a high-fat meal in Treatment Periods 2 through 4, respectively.
  Interventions: Drug: QRL-101
- Treatment Sequence 3 (Formulation 3, 1, and 2) (Experimental): Participants randomized to Treatment Sequence 3 will receive Formulation 3 in the fasted condition in Treatment Period 1, followed by Formulation 3, 1, and 2 in the presence of a high-fat meal in Treatment Periods 2 through 4, respectively.
  Interventions: Drug: QRL-101
- Treatment Sequence 4 (Formulation 2, 1, and 3) (Experimental): Participants randomized to Treatment Sequence 4 will receive Formulation 1 in the fasted condition in Treatment Period 1, followed by Formulation 1, 3, and 2 in the presence of a high-fat meal in Treatment Periods 2 through 4, respectively.
  Interventions: Drug: QRL-101
- Treatment Sequence 5 (Formulation 2, 1, and 3) (Experimental): Participants randomized to Treatment Sequence 5 will receive Formulation 2 in the fasted condition in Treatment Period 1, followed by Formulation 2, 1, and 3 in the presence of a high-fat meal in Treatment Periods 2 through 4, respectively.
  Interventions: Drug: QRL-101
- Treatment Sequence 6 (Formulation 3, 2, and 1) (Experimental): Participants randomized to Treatment Sequence 6 will receive Formulation 3 in the fasted condition in Treatment Period 1, followed by Formulation 3, 2, and 1 in the presence of a high-fat meal in Treatment Periods 2 through 4, respectively.
  Interventions: Drug: QRL-101

INTERVENTIONS:
Drug: QRL-101 — This cross-over design study will evaluate three formulations (Formulations 1, 2, and 3) of QRL-101, beginning in a fasted condition before moving to a fed cross-over design.

SUMMARY:
This study aims to evaluate the pharmacokinetics of three QRL-101 formulations in a fasted condition or in the presence of a high-fat meal in healthy participants.

DETAILED DESCRIPTION:
This is a randomized, open-label, single-dose, crossover study to evaluate the PK of three formulations of QRL-101 beginning in a fasted condition before moving to a fed cross-over design. Approximately 24 healthy participants will be enrolled in a 3-formulation, 4-period, 6-sequence crossover study design to evaluate the PK characteristics of three formulations of QRL-101.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years of age inclusive at the time of signing the informed consent.
2. Clinical chemistry laboratory values within acceptable range for the population, as per investigator judgment.
3. Body mass index of 18 to 32 kg/m2 (inclusive).
4. Willing and able to practice effective contraception.

Exclusion Criteria:

1. Currently enrolled in any other clinical trial involving a study drug or off-label use of a drug or device, or any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Any participant in >4 studies a year and/or has participated in a clinical trial within 1 month of the expected dosing date.
3. History or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric, or neurological disease, convulsions, or any clinically significant laboratory abnormality that, in the judgment of the investigator, indicate a medical problem that would preclude study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Plasma PK profile (AUCinf) | Baseline through Follow up (Day 9)
  The area under the curve to infinity
Plasma PK profile (AUClast) | Baseline through Follow up (Day 9)
  The area under the curve to the last measurable time point
Plasma PK profile (Cmax) | Baseline through Follow up (Day 9)
  Maximum concentration observed
Plasma PK profile (Ctrough) | Baseline through Follow up (Day 9)
  Trough level concentration for defined dose regimen
Plasma PK profile (Tmax) | Baseline through Follow up (Day 9)
  The time to peak drug concentration

SECONDARY OUTCOMES:
Safety and tolerability | Baseline through Follow up (Day 9)
  Adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Salah Hadi, MD, Principal Investigator — ICON plc
Locations (1):
- ICON plc. Van Swietenlaan 6, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No